CLINICAL TRIAL: NCT05209945
Title: High-Frequency Whole Body Vibration Activates Tonic Vibration Reflex
Brief Title: Whole Body Vibration and Tonic Vibration Reflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan KARACAN, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WBVTVR
Record Dates: First submitted 2022-01-03; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Vibration; Exposure; Muscle Physiology
Keywords: muscle strength; vibration; tonic vibration reflex
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibration (Experimental): Vibration (WBV, heel, and tendon vibration) was applied to participants
  Interventions: Procedure: vibration

INTERVENTIONS:
Procedure: vibration — whole-body vibration, heel and soleus tendon vibrations were applied to the human body

SUMMARY:
Whole-body vibration (WBV) has beneficial neuromuscular effects on muscle strength increase. Supraspinal, spinal, and peripheral mechanisms have been proposed to explain these beneficial effects. The most commonly proposed explanatory mechanism is spinal segmental reflexes. However, the neuronal circuit and receptors of the reflex response have not been defined precisely. A group of researchers found that the reflex system is the Tonic vibration reflex (TVR) under the neuromuscular effects of WBV; Other researchers claim that WBV activates a different spinal reflex than TVR. Tonic vibration reflex is a polysynaptic reflex that occurs as a result of muscle spindle activation, in which more than 100 Hz vibrations are applied to the belly or tendon of the muscle. A group of researchers argues that WBV activates the spinal reflex response, but this reflex response is different from TVR. According to them, WBV-induced reflex (WBV-IR) response latency is longer than TVR latency. WBV activates TVR at very attenuated amplitude; WBV activates a different spinal reflex with longer latency at medium and high amplitude vibration. They reported that although the H-reflex, T-reflex, and TVR latency was longer in the spastic soleus muscle than normotonic soleus muscle, where the muscle spindle and Ia afferent pathway were hyperactive. However, the WBV-IR latency was similar in both spastic and normotonic soleus muscle. According to our hypothesis, the reflex system activated by WBV changes depending on vibration frequency: if the high-frequency (100-150 Hz) WBV is applied, the tonic vibration reflex is activated; if the low-frequency (30-40 Hz) WBV is applied, the bone myoregulation reflex is activated. The purpose of this research is to test this hypothesis.

DETAILED DESCRIPTION:
Seven healthy recreationally active males between the ages of 26 and 35 volunteered to participate in this study. All subjects received pre-study informed consent. All experimental procedures were designed with the Helsinki declaration in mind and approved by the local ethics committee. All subjects performed a familiarization trial to acclimate subjects to the WBV stimulus. WBV-IR and TVR latency of soleus muscle were then measured in the quiet standing position. The vibrations (WBV or tendon) sequence were applied randomly to negate any order/time effect. The subject rested for five minutes between the WBV and tendon vibration. The WBV application was delivered using a PowerPlate Pro5 device (PowerPlate International, Amsterdam, The Netherlands). First, 30 Hz, low amplitude (1 mm) vibration with a duration of 30 seconds was applied to each subject for familiarization purposes. After three minutes of rest, low-amplitude (1 mm) WBV testing was performed in random order in quiet standing positions. In a WBV set, three different vibration frequencies (30, 35, and 40 Hz), each lasting for 30 s with 3-s rest intervals, were delivered. The local vibration was applied to the mid-point of the right Achilles tendon by using a custom-made vibrator. The head of the tendon vibrator was in light contact with the underlying skin. Tendon vibrations were applied by the same researcher. Three different vibration frequencies (100, 135, and 150 Hz) were delivered, lasting for 30 s with 3-s rest intervals. A local vibration was applied to the right heel using the same custom-made vibrator. Tendon vibrations were applied by the same researcher. Three different vibration frequencies (100, 135, and 150 Hz) were delivered, lasting for 30 s with 3-s rest intervals.

The surface electromyography (SEMG) recorded from the soleus and acceleration data were collected simultaneously using data acquisition and analysis system (PowerLab ® software, ADInstruments, Oxford, UK). Disposable self-adhesive bipolar Ag/AgCl (Covidien Kendall, Dublin, Ireland) surface electrodes were placed on the right soleus belly 4 cm apart. The skin overlying the muscle was shaved, light abrasion was applied, and the skin was cleaned with alcohol to reduce the skin resistance. To determine TVR latency, a light (2.9 g) piezoelectric accelerometer (LIS344ALH, ECOPACK®, Mansfield, TX, USA) was firmly fixed using adhesive tape on the skin overlying the right Achilles tendon. To determine WBV-IR latency, an identical accelerometer was firmly mounted on the WBV platform. The acceleration and SEMG signals were recorded at a sampling frequency of 20 kHz. Accelerometer recordings were filtered with a high-pass filter set at 5 Hz. SEMG data obtained during WBV were bandpass filtered at 80-500 Hz to reduce vibration-induced movement artifacts and then full-wave rectified. Similarly, SEMG data obtained during tendon vibration were bandpass filtered at 160-500 Hz and then full-wave rectified. WBV-IR and TVR latencies were then calculated by using the cumulative average method.

An electronic reflex hammer (Elcon, Germany) was used to determine T-reflex latency. All latencies were normalized to the body height of each participant.

Latency was expressed as milliseconds (ms).

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Being a young adult (20-45 years old)
* Volunteer

Exclusion Criteria:

* Scar, dermatitis, etc. in the skin tissue
* Kidney stone history
* Fracture in the lower extremity, history of orthopedic surgery
* Heart disease, Hypertension
* Dizziness
* Metabolic bone diseases, including osteoporosis
* History of bone occupying lesion, neoplasia, osteomyelitis
* Degenerative, inflammatory diseases of the joints of the lower extremities
* Lower extremity thrombophlebitis
* Lower extremity motor loss, sensory loss, muscle atrophy
* Subjects who cannot tolerate whole-body vibration

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
WBV-IR latency | during intervention, an average of 1 minute
  Whole-body vibration induced reflex latency
TVR latency | during intervention, an average of 1 minute
  Tonic vibration reflex latency
Heel vibration induced reflex latency | during intervention, an average of 1 minute
  Vibration was applied to the right heel. The reflex latency induced by the heel vibration was measured.
T-reflex latency | during intervention, an average of 1 minute
  Latency of the Achilles tendon reflex

CONTACTS AND LOCATIONS:
Overall Officials: İLHAN KARACAN, Study Chair — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)